CLINICAL TRIAL: NCT02235922
Title: Effects of a Dual Task Protocol on Cognition and Functionality in Non-sedentary Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Anielle C M Takahashi, principal investigator, Universidade Federal de Sao Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAPESI-01
Record Dates: First submitted 2014-09-06; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Non-sedentary
Keywords: Aged; Exercise; Cognition; Functional capacity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual task training (Experimental): Dual task training
  Interventions: Other: Dual task training
- Conventional training (Experimental): Conventional training
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: Dual task training — The dual task training consisted of individuals subjected to a multicomponent exercise program associated to cognitive tasks.
  Arms: Dual task training
Other: Conventional training — The conventional training consisted of individuals subjected to a multicomponent exercise program.
  Arms: Conventional training

SUMMARY:
The purpose of this study is to analyze the effects of a dual task protocol on cognitive domains and functional capacity in non-sedentary older adults.

The hypothesis of the present study is that older people undergoing to a dual task exercise protocol have greater benefits on cognition and functional performance, compared to a standard exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* aged over 60 years
* community people
* ability to walk alone
* non-sedentary

Exclusion Criteria:

* non-realization of any cognitive or functional assessment
* presence of Parkinson's Disease, Dementia and Stroke with motor sequel
* frequency to trainings below 70%

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes on cognition after 3 months of training | Assessed at baseline and after 3 months of training
  Cognition was assessed by Montreal Cognitive Assessment and Mini-Mental State Examination
Changes on functional capacity after 3 months of training | Assessed at baseline and after 3 months of training
  Functional capacity was assessed by Timed up and go test, Timed up and go test associated to a cognitive task and sit to stand test.

CONTACTS AND LOCATIONS:
Overall Officials: Anielle Takahashi, doctorate, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil